CLINICAL TRIAL: NCT07131540
Title: National Collaborative Centre for Hepatic Regenerative Medicine (NC-CHRM): To Study the Safety and Efficacy of Mesenchymal Stem-Cell Therapy in the Management of Non-viral ACLF Patients: Phase-I Clinical Study
Brief Title: National Collaborative Centre for Hepatic Regenerative Medicine (NC-CHRM): Phase I Study on Safety and Efficacy of Mesenchymal Stem-Cell (MSC) Therapy in Non-Viral Acute-on-Chronic Liver Failure (ACLF)
Acronym: NC-CHRM
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Collaborators: Indian Council of Medical Research (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-ACLF-70
Record Dates: First submitted 2025-07-11; First posted 2025-08-20 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Acute-On-Chronic Liver Failure
Keywords: ACLF; MSC; Liver failure
MeSH Terms: conditions — Acute-On-Chronic Liver Failure; Liver Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Safety and feasibility of ucMSCs therapy in non-viral ACLF (Phase-1) (Experimental): ACLF patients as per the definition of Asian Pacific association for the study of the liver (APASL) will be enrolled for safety and feasibility study of umbilical cord mesenchymal stem cells (ucMSCs). To test the safety and tolerability of ucMSC 1 million/kg will be given intra-venously once a week for 4 week in 10 ACLF patients. 250 ml normal saline will be infused 30 minutes prior to ucMSCs infusion. The fresh ucMSCs will be taken from ILBS cGMP facility and will be infused through IV canula peripherally over 30 minutes followed by a further 250 ml normal saline over 20-30 minutes. A baseline early warning score (EWS) will be undertaken with continuous monitoring of pulse and with blood pressure checks every 5 minutes during the cell infusion and then every 15 minutes during the subsequent 2-hour observation period, then every hour for the remaining 10-hour observation period (minimum total of 12 hours observation) after cell infusion.
  Interventions: Drug: umbilical cord Mesenchymal Stem Cell

INTERVENTIONS:
Drug: umbilical cord Mesenchymal Stem Cell — To test the safety and tolerability of ucMSC 1 million/kg will be given intra-venously once a week for 4 week in 10 ACLF patients. 250 ml normal saline will be infused 30 minutes prior to ucMSCs infusion. The fresh ucMSCs will be taken from ILBS cGMP facility and will be infused through IV canula peripherally over 30 minutes followed by a further 250 ml normal saline over 20-30 minutes.

SUMMARY:
Liver disease deaths are rising, but transplants remain scarce in India. With over 100,000 needed annually and only ~2,500 performed, non-transplant options are urgently needed. Regenerative therapy, especially MSCs, shows promise but lacks validation, particularly for non-viral Acute on Chronic Liver Failure (ACLF). The proposed NC-CHRM aims to develop and validate MSC-based therapy to promote native liver regeneration and offer a safe, effective, transplant-free treatment.

DETAILED DESCRIPTION:
The incidence of deaths from chronic liver diseases (CLD) and cirrhosis are rapidly increasing globally, including India. Liver transplant is the only curative option. Unfortunately, transplant is often not feasible. There is a need for nearly 100,000 liver transplants every year in India, though, only about 2,500 transplants are being done at present across the country. There is therefore, a huge unmet need of developing non-transplant options for chronic liver disease patients. In this regard emerging science of regenerative therapy holds great promises but therapeutic benefit of these therapies is limited due to lack of clinical validation.

Novelty: Liver failure is failure of regeneration hence, potentiating native liver repair and regeneration can serve as potential non-transplant approaches. Others and the investigators have shown in experimental studies that mesenchymal stem cells (MSCs) can improve hepatic regeneration. MSC therapy trials in decompensated cirrhosis and viral ACLF in Korea, China and Japan have shown promise but their utility in non-viral ACLF is limited. In the proposed National Collaborative Centre for Hepatic Regenerative Medicine (NC-CHRM) the investigators will use this novel regenerative medicine approaches MSC for management of acute liver failure in non-viral ACLF to develop safe and effective regenerative therapy clinical protocol for transplant free management of liver failure in cirrhosis. Using integrated cellular, molecular and functional analysis the investigators will also establish their mechanism of action and identify biomarker to access therapeutic response.

ELIGIBILITY:
Inclusion Criteria:

* ACLF patients with Model for End-Stage Liver Disease (MELD) >18 or APASL ACLF Research Consortium (AARC) grade 2 or more with (no or single extrahepatic organ dysfunction or failure having no option of liver transplant).

Exclusion Criteria:

* Age <18 or >65 yrs
* Patients with active sepsis
* Patients with hepatic venous outflow tract obstruction (HVOTO) or Extrahepatic portal vein obstruction (EHPVO)
* Hepatocellular carcinoma (beyond Milan) or any extrahepatic malignancy
* Active bleed (mucosal or variceal) or severe coagulopathy (platelets <20,000 or INR>4)
* Patients with refractory shock requiring norepinephrine >0.5ug/kg/min
* Patients with severe Acute Respiratory Distress Syndrome (ARDS) with Pa02/Fi02 <150
* Patients with retroviral infections
* Autoimmune hepatitis
* Viral etiology of liver disease
* Co-existent Hepatitis B, Hepatitis C, HIV
* Chronic kidney disease
* Multiorgan failure or disseminated intravascular coagulation (DIC)
* Patients improving on standard medical treatment
* Patients on immunosuppressive medications
* Pregnancy or active breastfeeding
* Known severe cardiopulmonary diseases (structural or valvular heart disease, coronary artery disease, coronary pulmonary disease, chronic kidney disease)
* Lack of informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2031-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Safety of ucMSC infusion in non-viral ACLF patients defined as proportion of patients completing the protocolized doses of MSC without major adverse effects requiring discontinuation. | Day 28 and Day 90

SECONDARY OUTCOMES:
Proportion of patients developing minor adverse effects | Day 28 and Day 90
Feasibility of ucMSC isolation and therapy Improvement in APASL ACLF Research Consortium (AARC) and MELD score from baseline at day 28 and day 90 | Day 28 and day 90
  Higher AARC (range: 5-15) and MELD (range: 6-40) scores indicate worse clinical status
Incidence of sepsis (assessed by positive culture reports) | Day 28 and Day 90
Incidence of renal dysfunction (evaluated by urine output and kidney function tests [KFTs]) | Day 28 and 90

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Shiv Kumar Sarin, DM, Principal Investigator — Institute of Liver & Biliary Sciences

IPD SHARING:
Plan to Share IPD: Undecided